CLINICAL TRIAL: NCT00647387
Title: Closure of Muscular Ventricular Septal Defects (VSDs) With the AMPLATZER Muscular VSD (MuVSD) Occluder - Post Approval Study
Acronym: VPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGA-016
Record Dates: First submitted 2008-03-27; First posted 2008-03-31 (Estimated); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ventricular Septal Defects
Keywords: muscular; ventricular; septal; defects; VSD
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Muscular VSD Occluder (Experimental): Implantation with the device
  Interventions: Device: Muscular VSD Occluder device implantation (AMPLATZER Muscular VSD Occluder)

INTERVENTIONS:
Device: Muscular VSD Occluder device implantation (AMPLATZER Muscular VSD Occluder) — Device

SUMMARY:
The AMPLATZER Muscular VSD Occluder was approved by the US Food and Drug Administration (FDA) in September, 2007. This study is designed to further evaluate the safety and effectiveness in subjects implanted with the AMPLATZER Muscular VSD Occluder.

ELIGIBILITY:
Inclusion Criteria:

1. complex congenital muscular ventricular septal defects (VSD) of significant size to warrant closure. Subjects must meet at least one of the following:

   1. Large volume left to right shunt (Qp/Qs >2:1),
   2. Pulmonary hypertension (PA pressure >50% systemic) and/or
   3. Clinical symptoms of congestive heart failure
   4. Banding of the pulmonary artery(ies) and in the opinion of the treating investigator closure of the VSD is clinically warranted.
2. Subjects must meet at least one of the following criteria to be considered high risk for standard transatrial or transarterial surgical closure based on anatomical conditions:

   1. Left ventriculotomy or an extensive right ventriculotomy,
   2. Failed previous VSD closure,
   3. Multiple apical and/or anterior muscular VSDs ("Swiss Cheese Septum"), and/or
   4. Posterior apical VSDs covered by trabeculae.
   5. Overall medical condition
3. Subject/legally authorized representative has signed the informed consent
4. Subject/legally authorized representative is willing to complete the follow-up requirements of this study

Exclusion Criteria:

1. Subjects with defects less than 4 mm distance from the semilunar (aortic and pulmonary) or atrioventricular valves (mitral and tricuspid)
2. Subjects with severely increased pulmonary vascular resistance above 7 Wood units and a right-to-left shunt and documented irreversible pulmonary vascular disease
3. Subjects with perimembranous (close to the aortic valve) VSD
4. Subjects with post-infarction VSD
5. Subjects who weigh < 5.2 kg
6. Subjects with sepsis (local/generalized)
7. Subjects with active bacterial infections
8. Subjects with contraindications to anti-platelets

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (48):
  - St. Joseph Hospital and Medical Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Arnold Palmer Hospital, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri-Kansas City School of Medicine, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Sunrise Hospital, Las Vegas, Nevada
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Children's Hospital of New York-Presbyterian, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist LeBonheur Healthcare, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - BC Children's Hospital, Vancouver, Bristish Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment began on 14 May 2008 and concluded on 24 February 2020. A total of 92 subjects were enrolled at 28 investigational sites in the United States and Canada. The post-approval requirements included subject follow-up through 5-years post-procedure.
Period: Overall Study
Arm/Group | Muscular VSD Occluder
Started | 92
Completed | 73
Not Completed | 19
Not completed — Lost to Follow-up | 6
Not completed — Unsuccessful implant | 5
Not completed — Device explanted | 3
Not completed — Other Reason | 3
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Analysis included prospectively (n=80) and retrospectively (n=12) enrolled subjects.
Arm/Group | Muscular VSD Occluder
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Ventricular septal defects (VSD) type [Count of Participants; unit: Participants]
  Single VSD | 45
  Multiple VSD | 32
  Swiss Cheese | 15

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness End Point: Technical Success
Description: Technical success was defined as successful deployment of the device (Amplatzer™ Muscular VSD Occluder) in subjects with the ventricular septal defect (VSD).
Time Frame: During the procedure
Population: The analysis population included all prospectively enrolled subjects only (N=80) who have an attempted device placement (defined as the delivery system enters the subject's body in an attempt to place a device), as retrospectively enrolled subjects were selected based on established Technical Success.
Measure: Count of Participants; unit: Participants
Arm/Group | Muscular VSD Occluder
Number analyzed (Participants) | 80
Participants | 75

2. Primary Outcome: Primary Effectiveness End Point: Acute Procedure Success
Description: Acute procedural success was defined as a defect with a ≤ 2mm residual shunt at the conclusion of the procedure, as reported by clinical sites.
Time Frame: At the end of the procedure
Population: The analysis population included all subjects who had an attempted device placement (defined as the delivery system enters the subject's body in an attempt to place a device).
Measure: Count of Participants; unit: Participants
Arm/Group | Muscular VSD Occluder
Number analyzed (Participants) | 91
Participants | 71

3. Primary Outcome: Primary Effectiveness End Point: Shunt Closure Success
Description: Subjects in whom a defect has ≤ 2 mm residual shunt at the 1-year follow-up visit (as evaluated by the independent echocardiography board).
Time Frame: 1-year follow-up visit
Population: The analysis of the shunt closure success included all enrolled subjects who had an attempted device placement (defined as the delivery system enters the subject's body in an attempt to place a device) and a 1-year follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Muscular VSD Occluder
Number analyzed (Participants) | 72
Participants | 68

4. Primary Outcome: Primary Safety Endpoint
Description: The proportion of subjects who experienced a serious adverse event (SAE) within 12 months of the procedure.
Time Frame: Within 12 months of the procedure
Population: The Primary Safety endpoint included all enrolled subjects except for withdrawn subjects with no adverse events within the first 12 months and consented screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Muscular VSD Occluder
Number analyzed (Participants) | 90
Participants | 47

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Muscular VSD Occluder
All-Cause Mortality (participants affected / at risk) | 2/92
Serious Adverse Events (participants affected / at risk) | 51/92
Other Adverse Events (participants affected / at risk) | 17/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Muscular VSD Occluder (N=92)
Abnormal Lab Value (Investigations) | 6
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Arterial Pulse Loss (Cardiac disorders) | 1
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (Respiratory, thoracic and mediastinal disorders) | 1
Asystole (Cardiac disorders) | 1
Ataxia (Nervous system disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Bacteremia (Infections and infestations) | 1
Bleeding (Blood and lymphatic system disorders) | 1
Blood Loss (Blood and lymphatic system disorders) | 3
Brain Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 2
Cardiac Arrest (Cardiac disorders) | 3
Cerebral Aneurysm (Nervous system disorders) | 1
Chronic Erosive Gastritis (Gastrointestinal disorders) | 1
Common Cold/Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1
Congestive Heart Failure (Cardiac disorders) | 3
Constipation (Metabolism and nutrition disorders) | 1
Cyanosis (Skin and subcutaneous tissue disorders) | 1
Dehydration (General disorders) | 2
Device Closure of ASD (Product Issues) | 3
Device Embolization (Product Issues) | 1
Device Malposition or Malfunction (Product Issues) | 1
Diarrhea (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
EKG Abnormalities (Investigations) | 1
Echo Finding (Investigations) | 1
Elective Cardiac Surgery (Cardiac disorders) | 13
Elective Procedure (Injury, poisoning and procedural complications) | 6
Elective Surgery (Surgical and medical procedures) | 4
Emesis/Vomiting (Gastrointestinal disorders) | 3
Failure to Thrive (General disorders) | 2
Febrile Seizures (General disorders) | 1
Fever (General disorders) | 3
Fracture (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1
Headache (General disorders) | 1
Heart Failure (Cardiac disorders) | 3
Hematemesis (Blood and lymphatic system disorders) | 1
Hemorrhage (Blood and lymphatic system disorders) | 1
Hypocalcemia (Blood and lymphatic system disorders) | 1
Hypotension (Blood and lymphatic system disorders) | 1
Intracerebral Haemorrhage (Vascular disorders) | 1
Intraventricular Haemorrhage (Vascular disorders) | 1
Ischemic Stroke (Vascular disorders) | 1
Junctional Escape Rhythm/Intermittent Junctional Rhythm (Cardiac disorders) | 1
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 1
PA Band Removal (Cardiac disorders) | 7
Partial Obstruction of the Aorta with a Gradient > 10mm Hg (Cardiac disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5
Poor Nutrition (Metabolism and nutrition disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Regurgitation/Pulmonary Insufficiency/Valvular Regurgitation: Pulmonary Valve (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Residual Shunt (Cardiac disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Syncytial Virus Infection (RSV) (Infections and infestations) | 2
Right Ventricular Outflow Tract (RVOT) Obstruction (Cardiac disorders) | 1
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 2
Sepsis (Infections and infestations) | 1
Septicemia (Infections and infestations) | 1
Stroke (Nervous system disorders) | 1
Systolic Dysfunction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1
Third Degree Heart Block (Complete Heart Block) (Cardiac disorders) | 1
Thrombus (Blood and lymphatic system disorders) | 3
Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation: Tricuspid Valve (Cardiac disorders) | 1
Urinary Tract Infections (Renal and urinary disorders) | 1
Viral Syndrome (Infections and infestations) | 1
Wound Dehiscence (Infections and infestations) | 1
Other (General disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Muscular VSD Occluder (N=92)
Arterial Hypertension/Hypertension (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Chest Pain (Cardiac disorders) | 2
Device Malposition or Malfunction (Product Issues) | 1
Diabetes Mellitus (Blood and lymphatic system disorders) | 1
Diastolic Dysfunction (Cardiac disorders) | 1
Elective Procedure (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
High Grade Block/Advanced AV Block (Cardiac disorders) | 1
Mobitz II Block (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Peripheral Arterial Occlusion (Cardiac disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Poor Nutrition (Metabolism and nutrition disorders) | 1
Pulmonary Vein Stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Seizure/Convulsions/Epilepsy (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation: Tricuspid Valve (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT00647387/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT00647387/SAP_001.pdf